CLINICAL TRIAL: NCT03704376
Title: Clinical Outcome Following Arthroscopic Knee Surgery (COFAKS)-Addendum
Brief Title: Clinical Comparison of Femoral Nerve Versus Adductor Canal Block Following Anterior Ligament Reconstruction
Acronym: FNB vs ACB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Hospital (Other)
Responsible Party: Principal Investigator, Lane Bailey, Director of Research and Education, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MH-14-0734 (addendum)
Record Dates: First submitted 2018-09-27; First posted 2018-10-12 (Actual); Results first posted 2018-12-11 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-09

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: Femoral Nerve Block; Adductor Canal Block
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Ropivacaine; Clonidine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Femoral Nerve Blockade (Active Comparator): Ultrasound guided FNB (30 ml of 0.2% ropivacaine with 100 mcg clonidine using a 22-gauge 40 mm ProBloc II insulated needle; Kimberly-Clark, Roswell, Georgia) below the inguinal ligament using a high-frequency linear ultrasound transducer (4-12 Hz; Mindray M7; Mindray North America, Mahwah, NJ) with stimulator confirmation.
  Interventions: Drug: 30 ml of 0.2% ropivacaine; Drug: 100 mcg clonidine; Device: High-frequency linear ultrasound transducer
- Adductor Canal Blockade (Active Comparator): Ultrasound guided ACB (15 ml of 0.2% ropivacaine with 100 mcg clonidine using a 22-gauge 40 mm ProBloc II insulated needle; Kimberly-Clark, Roswell, Georgia) at the mid-thigh using a high-frequency linear ultrasound transducer (4-12 Hz; Mindray M7; Mindray North America, Mahwah, NJ).
  Interventions: Drug: 15 ml of 0.2% ropivacaine; Drug: 100 mcg clonidine; Device: High-frequency linear ultrasound transducer

INTERVENTIONS:
Drug: 30 ml of 0.2% ropivacaine
  Arms: Femoral Nerve Blockade
Drug: 15 ml of 0.2% ropivacaine
  Arms: Adductor Canal Blockade
Drug: 100 mcg clonidine
Device: High-frequency linear ultrasound transducer

SUMMARY:
This study will examine the potential differences between femoral nerve blockade (FNB) and adductor canal blockade (ACB) for pain control and quadriceps muscle activation for patients following anterior cruciate ligament (ACL) reconstruction.

DETAILED DESCRIPTION:
Adequate pain control following anterior cruciate ligament reconstruction (ACL) often requires a regional nerve block. The femoral nerve block (FNB) has been traditionally employed. More recently, ultrasound application to regional nerve blocks allows for the use of alternatives such as the adductor canal block following ACL reconstruction. In 2009, Manickam et al. were the first to describe the ultrasound guided adductor canal technique for the purposes of knee joint analgesia. Unlike other traditional techniques that seek to cause a sensory as well as a motor blockade, the adductor canal block attempts to spare the motor block of the neighboring distributions in an attempt to offer selective analgesia and strength preservation. Chisholm et al demonstrated the adductor canal block provides similar and adequate postoperative analgesia when compared to the FNB, following arthroscopic ACL reconstruction with patellar tendon autograft. Their study focused on analgesia and did not evaluate quadriceps function or impact on rehabilitation. Sharma et al drew the first association between femoral nerve blocks and increased fall risk due to muscle weakness in total knee arthroplasty population. A randomized, blinded study to compare quadriceps strength following adductor canal versus FNB was performed by Kwofie et al. They showed that compared with FNB, adductor canal block results in significant quadriceps motor sparing and significantly preserved balance. These studies focused on acute muscle weakness after regional anesthesia and its relation to safety. Quadriceps function is very important in rehabilitation of ACL reconstruction. Luo et al demonstrated long term deficits related to FNB. They demonstrated that patients treated with FNB after ACL reconstruction had significant isokinetic deficits in knee extension and flexion strength at 6 months when compared with patients who did not receive a nerve block. Patients without a block were 4 times more likely to meet criteria for clearance to return to sports at 6 months. In addition, Krych et al found significantly inferior quadriceps strength and function at 6 months in FNB group. Based on the available literature, we aim to compare femoral nerve versus adductor canal block in regards to pain control and muscle strength in ACL reconstruction patients until return to sport.

ELIGIBILITY:
Inclusion Criteria:

* Males & Females ages 16-30 yrs
* Undergoing ACL reconstruction by Co-Investigator (Walter Lowe)
* Receiving peri-operative FNB or ACB

Exclusion Criteria:

* Not enrolled within the COFAKS study
* Receiving intrathecal nerve blockade or no blockade

Ages: 16 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-11-16 (Actual); Study Completion 2017-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lane Bailey, PhD, PT, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center-Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duncan BR, Reid M, Kleihege J, Higbie S, Gardner EP, Lowe W, Bailey L. Comparison of Psychological Readiness to Return to Sport After Primary Versus Revision Anterior Cruciate Ligament Reconstruction. Orthop J Sports Med. 2023 May 2;11(5):23259671231159408. doi: 10.1177/23259671231159408. eCollection 2023 May. PMID 37152546
- [Derived] Galloway C, Ward H, Higbie S, Kleihege J, Kumaravel M, Lowe WR, Bailey L. Relationship Between Bone Bruise Volume and Patient Outcomes After ACL Reconstruction. Orthop J Sports Med. 2023 Feb 24;11(2):23259671221146205. doi: 10.1177/23259671221146205. eCollection 2023 Feb. PMID 36860772
- [Derived] Bailey L, Weldon M, Kleihege J, Lauck K, Syed M, Mascarenhas R, Lowe WR. Platelet-Rich Plasma Augmentation of Meniscal Repair in the Setting of Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2021 Oct;49(12):3287-3292. doi: 10.1177/03635465211036471. Epub 2021 Sep 3. PMID 34477016
- [Derived] Worsham J, Lowe WR, Copa D, Williams S, Kleihege J, Lauck K, Mascarenhas R, Bailey L. Subsequent Surgery for Loss of Motion After Anterior Cruciate Ligament Reconstruction Does Not Influence Function at 2 Years: A Matched Case-Control Analysis. Am J Sports Med. 2019 Sep;47(11):2550-2556. doi: 10.1177/0363546519863347. Epub 2019 Jul 26. PMID 31348866
- [Derived] Bailey L, Griffin J, Elliott M, Wu J, Papavasiliou T, Harner C, Lowe W. Adductor Canal Nerve Versus Femoral Nerve Blockade for Pain Control and Quadriceps Function Following Anterior Cruciate Ligament Reconstruction With Patellar Tendon Autograft: A Prospective Randomized Trial. Arthroscopy. 2019 Mar;35(3):921-929. doi: 10.1016/j.arthro.2018.10.149. Epub 2019 Feb 4. PMID 30733025

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 125 were enrolled, but 39 were excluded because they ended up receiving a different type of graft.
Groups:
- Femoral Nerve Blockade: Ultrasound guided FNB (30 ml of 0.2% ropivacaine with 100 mcg clonidine using a 22-gauge 40 mm ProBloc II insulated needle; Kimberly-Clark, Roswell, Georgia) below the inguinal ligament using a high-frequency linear ultrasound transducer (4-12 Hz; Mindray M7; Mindray North America, Mahwah, NJ) with stimulator confirmation.
  30 ml of 0.2% ropivacaine
  100 mcg clonidine
  High-frequency linear ultrasound transducer
- Adductor Canal Blockade: Ultrasound guided ACB (15 ml of 0.2% ropivacaine with 100 mcg clonidine using a 22-gauge 40 mm ProBloc II insulated needle; Kimberly-Clark, Roswell, Georgia) at the mid-thigh using a high-frequency linear ultrasound transducer (4-12 Hz; Mindray M7; Mindray North America, Mahwah, NJ).
  15 ml of 0.2% ropivacaine
  100 mcg clonidine
  High-frequency linear ultrasound transducer
Period: Overall Study
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Started | 42 | 44
Completed | 38 | 40
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade | Total
Number analyzed (Participants) | 38 | 40 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (8.8) | 21.0 (7.3) | 22.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 20 | 23 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Quadriceps Muscle Activation as Assessed by Surface Electromyography (sEMG)
Description: Quadriceps muscle activation was examined using surface electromyography (sEMG) of the vastus medialis oblique muscle. Peak sEMG activity was recorded in microvolts (uV) on the surgical and contralateral limbs while performing five maximal effort isometric contractions in full knee extension--the reported values are equal to the quadriceps sEMG in uV of the contralateral limb minus the quadriceps sEMG in uV of the surgical limb.
Time Frame: Post-operative day 1
Measure: Mean (Standard Deviation); unit: microvolts (uV)
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
microvolts (uV) | 266.5 (52.4) | 212.5 (65.1)

2. Primary Outcome: Quadriceps Muscle Activation as Assessed by Surface Electromyography (EMG)
Description: as for outcome 1
Time Frame: Post-operative day 14
Measure: Mean (Standard Deviation); unit: microvolts (uV)
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
microvolts (uV) | 183.2 (41.8) | 126.5 (48.9)

3. Primary Outcome: Quadriceps Muscle Activation as Assessed by Surface Electromyography (EMG)
Description: as for outcome 1
Time Frame: 4 weeks post operative
Measure: Mean (Standard Deviation); unit: microvolts (uV)
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
microvolts (uV) | 109.1 (32.2) | 94.1 (33.2)

4. Secondary Outcome: Number of Successful Repetitions With Straight Leg Raise Test
Description: The straight leg raise assessment was performed in a standardized long-sitting position with well-knee flexed to 90 degrees. Patients were asked to complete 30 repetitions of straight leg raises with a small bolster supporting the heel using the following criteria; (1) perform with no visible quad lag (2) reach the height of the opposite tibial tubercle and (3) maintain a controlled rate of 30 hertz for the ascending and descending phases. The examination was only performed on the surgical limb and the absolute number of successful repetitions is reported.
Time Frame: Post-operative day 1
Measure: Mean (Standard Deviation); unit: number of repetitions
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
number of repetitions | 3.2 (6.1) | 6.2 (8.0)

5. Secondary Outcome: Number of Successful Repetitions With Straight Leg Raise Test
Description: as for outcome 4
Time Frame: Post-operative day 14
Measure: Mean (Standard Deviation); unit: number of repetitions
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
number of repetitions | 23.3 (10.6) | 24.2 (10.9)

6. Secondary Outcome: Number of Successful Repetitions With Straight Leg Raise Test
Description: as for outcome 4
Time Frame: 4 weeks post operative
Measure: Mean (Standard Deviation); unit: number of repetitions
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
number of repetitions | 29.7 (1.4) | 30 (0.0)

7. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, 0 being the better outcome.
Time Frame: 1 hr post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
units on a scale | 0.81 (2.09) | 0.8 (2.23)

8. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better outcome.
Time Frame: 2 hr post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
units on a scale | 1.78 (2.61) | 2.13 (3.2)

9. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better
Time Frame: 3 hr post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
units on a scale | 2.65 (2.8) | 3.23 (3.3)

10. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better outcome.
Time Frame: 4 hr post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
units on a scale | 2.83 (2.6) | 2.87 (3.08)

11. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better outcome.
Time Frame: 5 hr post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
units on a scale | 2.97 (2.47) | 3.06 (2.94)

12. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better outcome.
Time Frame: 6 hr post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
units on a scale | 2.63 (2.51) | 3.03 (2.99)

13. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better outcome.
Time Frame: 7 hr post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
units on a scale | 2.83 (2.22) | 2.81 (2.63)

14. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better outcome.
Time Frame: 8 hr post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
units on a scale | 2.84 (2.04) | 2.57 (2.63)

15. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better outcome.
Time Frame: 9 hr post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
units on a scale | 2.91 (2.07) | 2.41 (2.27)

16. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better outcome.
Time Frame: 10 hr post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
units on a scale | 2 (1.9) | 2.53 (1.89)

17. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better outcome.
Time Frame: 11 hr post surgery
Population: No participants were analyzed for this time point because participants were discharged from hospital at around 10 hours, before this time point would have occurred.
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better outcome.
Time Frame: 12 hr post surgery
Population: as for outcome 17
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Postoperative Pain Control as Assessed by a Numeric Pain Rating Scale
Description: The items are scored on a visual analogical scale from 0-10, with 0 being the better
Time Frame: Postoperative physicians visit
Population: Patients were not analyzed at postoperative physicians visit.
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Narcotics Use as Assessed by Morphine Equivalents Consumed
Description: morphine equivalents consumed during the entire post-anesthesia care unit (PACU) visit post surgery will be obtained from the All-scripts electronic medical record (EMR) system.
Time Frame: Entire post-anesthesia care unit (PACU) visit post surgery, PACU range 1 hr to 12 hrs post surgery
Measure: Mean (Standard Deviation); unit: milligrams (mg)
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
Number analyzed (Participants) | 38 | 40
milligrams (mg) | 14.8 (8.3) | 16.0 (7.4)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Femoral Nerve Blockade | Adductor Canal Blockade
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/40
Other Adverse Events (participants affected / at risk) | 16/38 | 11/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Femoral Nerve Blockade (N=38) | Adductor Canal Blockade (N=40)
Anterior Knee Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (8)
Knee Extension Loss (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Reinjury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-02): https://cdn.clinicaltrials.gov/large-docs/76/NCT03704376/Prot_SAP_000.pdf